CLINICAL TRIAL: NCT01042990
Title: Testing Adaptive Physical Activity in Stroke
Acronym: TAPAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Baltimore VA Medical Center (U.S. Federal Agency)
Collaborators: University of Maryland (Other)
Responsible Party: Richard F. Macko, University of Maryland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HP-00040264
Record Dates: First submitted 2010-01-05; First posted 2010-01-06 (Estimated); Last update posted 2010-01-06 (Estimated); Status verified 2009-12

CONDITIONS: Stroke
Keywords: Stroke; Exercise; Balance; Dynamic Gait; Cardiovascular Fitness
MeSH Terms: conditions — Stroke; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Home Exercise Only (Active Comparator): Participants receive education and instruction on a home exercise program which they do on their own, with intermittent encouragement from study personnel.
  Interventions: Other: Adaptive Physical Activity
- APA (Experimental): Participants exercise in a gym setting 3x/week for six months, performing gait and balance exercises along with a progressive walking program.
  Interventions: Other: Adaptive Physical Activity
- APA+TM (Experimental): Participants exercise in a gym setting 3x/week for six months, performing a combined program of adaptive physical activity (gait and balance training) and progressive treadmill walking.
  Interventions: Other: Adaptive Physical Activity

INTERVENTIONS:
Other: Adaptive Physical Activity — Structured gait, balance, and progressive walking program performed in a group gym setting 3x/week for 6 months

SUMMARY:
"Testing Adaptive Physical Activity in Stroke" tests the idea that adaptive physical activity (APA) will improve fitness, balance and walking function, daily step activity, and outcomes related to quality of life in individuals with chronic stroke. Adaptive physical activity is an exercise model that combines aerobic exercise with balance and gait training in a socially reinforcing group setting. Individualized homework assignments encourage integration of exercise into daily life routines. Our specific aims are:

1. to determine whether APA improves cardiovascular fitness and metabolic health
2. to measure the effects of APA on gait and balance, ambulatory activity, and ADL function
3. to determine whether APA affects self-reported outcomes related to self-efficacy, fatigue, and stroke-specific quality of life

ELIGIBILITY:
Inclusion Criteria:

1. Ischemic stroke greater than or equal to 6 months prior in men or women ages 40- or older. Hemorrhagic stroke greater than or equal to one year prior in men or women ages 40-or older.
2. Residual hemiparetic gait deficits.
3. Already completed all conventional inpatient and outpatient physical therapy.
4. Adequate language and neurocognitive function to participate in exercise testing and training (specific screening instruments used.)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2008-09; Primary Completion 2011-09 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
VO2 Peak | baseline, 3 months, 6 months, and 3 months post-intervention
Berg Balance Scale | baseline, 3 months, 6 months, and 3 months post-intervention
Dynamic Gait Index | Baseline, 3 months, 6 months, and 3 months post intervention
Step Activity Monitoring | Baseline, 3 months, 6 months, and 3 months post-intervention
6 Minute Walks | Baseline, 3 months, 6 months, and 3 months post-intervention

SECONDARY OUTCOMES:
Psychosocial questionnaires | baseline, 3 months, 6 months, and 3 months post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Richard F Macko, MD, Principal Investigator — University of Maryland; Kathleen M Michael, PhD, Principal Investigator — University of Maryland; Andrew P Goldberg, MD, Principal Investigator — University of Maryland
Locations (1):
- Baltimore VAMC, Baltimore, Maryland, United States

REFERENCES:
- [Result] Michael K, Goldberg AP, Treuth MS, Beans J, Normandt P, Macko RF. Progressive adaptive physical activity in stroke improves balance, gait, and fitness: preliminary results. Top Stroke Rehabil. 2009 Mar-Apr;16(2):133-9. doi: 10.1310/tsr1602-133. PMID 19581199